CLINICAL TRIAL: NCT01944137
Title: Improving Care After Chemotherapy
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lara Traeger, Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-258
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Non-small Cell Lung Cancer; Colorectal Cancer; Breast Cancer
Keywords: colonic neoplasms; Lung neoplasms; patient-centered nursing; breast neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Participant will receive standard cancer care
- Nursing Intervention (Experimental): Participants will receive 4 planned phone calls from nurse practitioners during their first 2 cycles of chemotherapy
  Interventions: Other: Nursing Intervention

INTERVENTIONS:
Other: Nursing Intervention — Participants will receive 4 planned phone calls from nurse practitioners during their first 2 cycles of chemotherapy, in order to proactively monitor and address chemotherapy-related symptoms.
  Arms: Nursing Intervention

SUMMARY:
The main purpose of this study is to examine changes in patient-reported symptoms during the first two cycles of neoadjuvant or adjuvant chemotherapy for non-small cell lung cancer (NSCLC), colorectal cancer (CRC) and breast cancer, among patients who receive standard care plus a proactive nursing intervention relative to patients who receive standard care alone. Interventions to improve symptom management and prevent urgent care needs in both the clinic and hospital for patients receiving chemotherapy with curative intent are needed to enhance the quality of cancer care.

DETAILED DESCRIPTION:
* Participants with NSCLC, CRC or breast cancer undergoing neoadjuvant or adjuvant chemotherapy will be asked to fill out self-report questionnaires at their first chemotherapy administration visit, in order to measure patient-reported symptoms, psychological distress, and satisfaction with oncology care.
* Participants will then be randomized into one of the two study groups: standard care with proactive phone calls from nurse practitioners or standard care alone.
* Participants assigned to the standard care group will be treated by their care team as would any other cancer patient.
* Participants assigned to the intervention group will receive four proactive phone calls from nurse practitioners designed to discuss symptom burden and management. Proactive phone calls will occur 2-4 days after chemotherapy administration and 5-7 days after chemotherapy administration, during cycles 1 and 2.
* Participants will be asked to fill out the same set of questionnaires during their second and third chemotherapy administration visits, to assess patient-reported symptoms, psychological distress, and satisfaction with oncology care.
* Medical records will be reviewed at 24-weeks following the first chemotherapy administration visit, to evaluate frequency of urgent outpatient cancer center visits, emergency department visits, and hospital admissions that occurred during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 or older)
* Newly diagnosed stage I-III colorectal cancer, non-small-cell lung cancer, or breast cancer
* Scheduled to receive neoadjuvant chemotherapy (i.e. pre-surgical cancer-directed therapy with curative intent) or adjuvant chemotherapy (i.e. post-surgical cancer-directed therapy with curative intent)
* Able to respond to questions in English

Exclusion Criteria:

* Already received 1 or more cycles of chemotherapy for the current regimen
* Unwilling or unable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline (i.e. first chemotherapy administration visit) in patient-reported symptoms as measured by the Memorial Symptom Assessment Scale-Short Form. | At approximately 2-3 weeks and 4-6 weeks post-baseline
  Eight symptom items assessing presence and level of distress per symptom over past week on a 5-point Likert type scale

SECONDARY OUTCOMES:
Change from baseline (i.e. first chemotherapy administration visit) in patient-reported psychological distress as measured by the Patient Health Questionnaire-4. | Approximately 2-3 weeks and 4-6 weeks post-baseline
  4-item screen of depression and anxiety symptoms
Change from baseline (i.e. first chemotherapy administration visit) in patient-reported satisfaction with oncology care as measured by the Family Caregiver Satisfaction-patient scale | Approximately 2-3 weeks and 4-6 weeks post-baseline
  13 items assess patient satisfaction with medical care on a 5-point Likert-type scale
Frequency of urgent outpatient Cancer Center visits, emergency department visits, and hospital admissions during six months post-baseline | Approximately six months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Theresa McDonnell, ACNP-BC, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States